CLINICAL TRIAL: NCT03871439
Title: A PHASE 1, OPEN LABEL, TWO-PERIOD, RANDOMIZED CROSSOVER STUDY TO COMPARE THE PHARMACOKINETICS OF TWO DIFFERENT FORMULATIONS OF PF-05221304 ADMINISTERED ORALLY TO HEALTHY ADULT SUBJECTS
Brief Title: OPEN LABEL, 2-PERIOD STUDY, TO COMPARE BIO-AVAILABILITY OF 2 DIFFERENT FORMULATIONS OF PF-05221304 IN HEALTHY ADULTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C1171007
Record Dates: First submitted 2019-02-25; First posted 2019-03-12 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-05221304 Formulation A (Experimental)
  Interventions: Drug: PF-05221304 Formulation A
- PF-05221304 Formulation B (Experimental)
  Interventions: Drug: PF-05221304 Formulation B

INTERVENTIONS:
Drug: PF-05221304 Formulation A — 50mg
  Arms: PF-05221304 Formulation A
Drug: PF-05221304 Formulation B — 50mg
  Arms: PF-05221304 Formulation B

SUMMARY:
The purpose of this study is to characterize the plasma pharmacokinetics of two formulations of PF 05221304 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18 and 55 years old inclusive
* Body Mass Index (BMI) of >= 17.5 and <= 30.4 kg/m2
* Total body weight > 50 kg (110lb)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, allergic disease or clinical findings

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Plasma PF-05221304 AUClast | Thirteen timepoints between 0-72 Hours
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Plasma PF-05221304 Cmax | Thirteen timepoints between 0-72 Hours
  Maximum Observed Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Number of Subjects Experiencing an Adverse Event | Up to 10 weeks from screening
  Number of Participants With Adverse Events (AEs) by Seriousness and Relationship to Treatment
Number of Participants With Clinical Laboratory Abnormalities | Up to 10 weeks from screening
  Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, lactate dehydrogenase, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, phosphate, bicarbonate); clinical chemistry (glucose, creatine kinase); immunology (CRP); urinalysis (dipstick [urine specific gravity, decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, bilirubin], microscopy [urine RBC, WBC, urate crystals, calcium, oxalate, miscellaneous [urine mucus and leucocytes]).
Number of Participants With Categorical Vital Signs Data | Up to 10 weeks from screening
  Number of participants with maximum increase from Baseline in sitting Systolic Blood Pressure and Diastolic Blood Pressure of greater than or equal to 30 mmHg
Number of Participants With Abnormal Electrocardiogram (ECG) | Up to 10 weeks from screening
  Criteria for potential clinical concern in ECG parameters: Maximum corrected QT interval (QTc) in range of 450 to less than 480 millisecond (msec), Maximum QTcB interval (Bazett's Correction) (msec) in range of 450 to less than 480 msec, Maximum QTcF interval (Fridericia's Correction) in range of 450 to less than 480 msec, maximum QTc interval increase from baseline in range of 30 to less than 60 msec and >=60 msec.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1171007